CLINICAL TRIAL: NCT00539539
Title: Controlled Study of the Clinical Effectiveness of Automated Real-Time Feedback on CPR Process Conducted at a Subset of ROC Sites
Brief Title: Automated Real-time Feedback on CPR Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); The Institute of Circulatory and Respiratory Health (ICRH) (Unknown); Defence Research and Development Canada (Industry)
Responsible Party: Principal Investigator, Susanne May, Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 30707-A; 5U01HL077863-08 (NIH); 28765 (Other: UW Human Subjects Division)
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2012-06-25 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-05

CONDITIONS: Heart Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Feedback On (Active Comparator): Automated real-time feedback on CPR Process activated
  Interventions: Other: Laerdal Q-CPR /technology
- Feedback Off (No Intervention): For the first three to six months, participating EMS agencies will have defibrillators with automated, real-time feedback inactivated. During this period, the baseline rate of ROSC (and secondary outcomes) will be collected. At the end of this baseline period, EMS agencies will be randomized to one of two interventions, with randomization stratified within site by agency, station, or device. All clusters will cross-over to the opposite feedback strategy at least once during the intervention phase.

INTERVENTIONS:
Other: Laerdal Q-CPR /technology — For the first three to six months, participating EMS agencies will have defibrillators with automated, real-time feedback inactivated. During this period, the baseline rate of ROSC (and secondary outcomes) will be collected. At the end of this baseline period, EMS agencies will be randomized to one of two interventions, with randomization stratified within site by agency, station, or device. All clusters will cross-over to the opposite feedback strategy at least once during the intervention phase.
  Arms: Feedback On

SUMMARY:
The purpose of this study is to evaluate whether or not real-time feedback on CPR process variables will increase rates of restoration of spontaneous circulation during prehospital resuscitation and upon arrival at the receiving emergency room as well as increase rates of survival to hospital discharge.

DETAILED DESCRIPTION:
A subset of emergency medical services (EMS) agencies that are participating in the Resuscitation Outcomes Consortium (ROC) are adopting new monitor/defibrillators that are capable of monitoring CPR process during attempted resuscitation of patients in cardiac arrest, as well as providing automated real-time feedback about this process to EMS providers so as to improve compliance with recommended guidelines for CPR. Monitoring of CPR process during attempted resuscitation is an important step towards reducing the potential for poorly-performed CPR to modify the effect of the study interventions upon outcome. Clusters formed of rigs, an individual agency or groups of agencies were randomized to turn feedback on or off. After a fixed period of time, each cluster crossed over to the other arm. An unequal number of subjects were enrolled during each period.

ELIGIBILITY:
Inclusion Criteria:

* all individuals who experience cardiac arrest outside the hospital,
* are evaluated by organized EMS personnel and: a) receive attempts at external defibrillation (by lay responders or emergency personnel) or receive chest compressions by organized EMS personnel.

Exclusion Criteria:

* Use of a mechanical CPR device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1586 (Actual)
Dates: Start 2007-02; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne May, PhD, Principal Investigator — University of Washington; Judy Powell, BSN, Study Director — University of Washington
Locations (3):
- United States (2):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington
- The Ottawa Hospital, Thunder Bay, Ontario, Canada

REFERENCES:
- [Derived] Hostler D, Everson-Stewart S, Rea TD, Stiell IG, Callaway CW, Kudenchuk PJ, Sears GK, Emerson SS, Nichol G; Resuscitation Outcomes Consortium Investigators. Effect of real-time feedback during cardiopulmonary resuscitation outside hospital: prospective, cluster-randomised trial. BMJ. 2011 Feb 4;342:d512. doi: 10.1136/bmj.d512. PMID 21296838
- See also: Click here for more information about this study: CPR Feedback Study — https://www.uwctc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Feedback On | Feedback Off
Started | 815 | 771
Completed | 815 | 771
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Feedback On | Feedback Off | Total
Number analyzed (Participants) | 815 | 771 | 1586
Age Categorical [Number; unit: participants] — Age is available on 1171 participants; 585 on feedback on arm; 586 on the feedback off arm
  participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 275 | 288 | 563
    >=65 years | 310 | 298 | 608
Age Continuous [Mean (Standard Deviation); unit: years] — Age available for 1171 participants; 585 on feedback arm; 586 on feedback off arm
  years | 65 (17) | 66 (17) | 66 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 295 | 291 | 586
  Male | 520 | 480 | 1000
Region of Enrollment [Number; unit: participants]
  United States | 777 | 766 | 1543
  Canada | 38 | 5 | 43

OUTCOME MEASURES:

1. Primary Outcome: Rate of ROSC During the Prehospital Resuscitation
Description: Return of spontaneous circulation (ROSC)
Time Frame: Prehospital resuscitation
Population: Intent to treat
Measure: Number; unit: Participants
Arm/Group | Feedback On | Feedback Off
Number analyzed (Participants) | 815 | 771
Participants | 361 | 345
Statistical Analysis 1: Comparison: Feedback On vs Feedback Off; Average change in cluster-specific rates of ROSC; Test type: Superiority or Other; p = 0.96, t-test, 2 sided; Risk Difference (RD) = 0.001, 95% CI 2-sided [-0.04 to 0.05]

2. Secondary Outcome: Pulses Present at ED Arrival.
Time Frame: Resuscitation
Population: Intention to treat. Presence of pulses not known for one participant on the feedback off arm. Analysis includes 815 participants on the feedback on arm and 770 on the feedback off arm.
Measure: Number; unit: Participants
Arm/Group | Feedback On | Feedback Off
Number analyzed (Participants) | 815 | 771
Participants | 260 | 243
Statistical Analysis 1: Comparison: Feedback On vs Feedback Off; Average difference in cluster-specific rates; Test type: Superiority or Other; p = 0.71, t-test, 2 sided; Risk Difference (RD) = -0.8, 95% CI 2-sided [-4.9 to 3.4]

3. Secondary Outcome: Survival to Hospital Discharge
Description: Survival to hospital discharge
Time Frame: Length of Hospitalization
Population: Intention to treat, with survival to hospital discharge missing for one participant on the feedback off arm. Analysis included 815 participants on the feedback on arm, and 770 on the feedback off arm.
Measure: Number; unit: Participants
Arm/Group | Feedback On | Feedback Off
Number analyzed (Participants) | 815 | 771
Participants | 92 | 96
Statistical Analysis 1: Comparison: Feedback On vs Feedback Off; Average change in cluster-specific risk difference; Test type: Superiority or Other; p = 0.21, t-test, 2 sided; By-cluster difference in outcome rates; Risk Difference (RD) = -0.015, 95% CI 2-sided [-0.039 to 0.009]

4. Secondary Outcome: CPR Fraction
Description: Percentage of time during CPR spend doing compressions.
Time Frame: Up to 10 minutes of CPR
Population: Intention to treat, with CPR fraction available for 604 participants on the feedback on arm, and 570 on the feedback off arm.
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Feedback On | Feedback Off
Number analyzed (Participants) | 815 | 771
Percentage | 66 (1) | 64 (1)
Statistical Analysis 1: Comparison: Feedback On vs Feedback Off; Cluster adjusted difference in average CPR fraction; Test type: Superiority or Other; p = 0.016, Regression, Linear; Difference in means, adjusted for cluster; Mean Difference (Net) = 1.9, 95% CI 2-sided [0.4 to 3.4]

5. Secondary Outcome: Compression Depth
Description: Average compression depth (mm) during the first 10 minutes of CPR.
Time Frame: Up to 10 minutes of CPR
Population: Intention to treat. Compression depth available for 529 participants on the feedback on arm and 467 on the feedback off arm.
Measure: Mean (Standard Error); unit: mm
Arm/Group | Feedback On | Feedback Off
Number analyzed (Participants) | 815 | 771
mm | 39.6 (0.4) | 37.8 (0.4)
Statistical Analysis 1: Comparison: Feedback On vs Feedback Off; Cluster adjusted difference in means; Test type: Superiority or Other; p = 0.005, Regression, Linear; Adjusted for randomization by cluster; Mean Difference (Net) = 1.6, 95% CI 2-sided [0.5 to 2.7]

6. Secondary Outcome: Compression Rate
Description: Average compression rate during the first 10 minutes of CPR.
Time Frame: Up to 10 minutes of CPR
Population: Intention to treat. Average compression rate available for 604 participants on the feedback on arm and 570 on the feedback off arm.
Measure: Mean (Standard Error); unit: Compressions per minute
Arm/Group | Feedback On | Feedback Off
Number analyzed (Participants) | 815 | 771
Compressions per minute | 103.1 (0.5) | 108.0 (0.7)
Statistical Analysis 1: Comparison: Feedback On vs Feedback Off; Cluster adjusted difference in average compression rate; Test type: Superiority or Other; p < 0.001, Regression, Linear; Mean Difference (Net) = -4.7, 95% CI 2-sided [-6.4 to -3.0]

7. Secondary Outcome: Percentage of Compressions With an Incomplete Release
Description: Percentage of compressions with incomplete release during the first ten minutes of CPR.
Time Frame: Up to 10 minutes of CPR
Population: Intention to treat. Incomplete release available for 529 participants on the feedback on arm and 467 on the feedback off arm.
Measure: Mean (Standard Error); unit: % of compressions w/ incomplete release
Arm/Group | Feedback On | Feedback Off
Number analyzed (Participants) | 815 | 771
% of compressions w/ incomplete release | 10.4 (1) | 14.6 (1)
Statistical Analysis 1: Comparison: Feedback On vs Feedback Off; Cluster adjusted difference in the average rate; Test type: Superiority or Other; p < 0.001, Regression, Linear; Mean Difference (Net) = -3.4, 95% CI 2-sided [-5.2 to -1.5]

8. Secondary Outcome: Ventilation Rate
Description: Average ventilation rate (breaths/minute) during the first ten minutes of CPR.
Time Frame: Up to 10 minutes of CPR
Population: Intention to treat. Ventilation rate available in 347 participants on the feedback on arm and 346 on the feedback off arm.
Measure: Mean (Standard Error); unit: breaths per minute
Arm/Group | Feedback On | Feedback Off
Number analyzed (Participants) | 815 | 771
breaths per minute | 5.8 (0.2) | 5.6 (0.2)
Statistical Analysis 1: Comparison: Feedback On vs Feedback Off; Cluster adjusted difference in average rate; Test type: Superiority or Other; p = 0.73, Regression, Linear; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.5 to 0.7]

ADVERSE EVENTS:
Time Frame: Pre-hospital resuscitation and hospitalization.
Arm/Group | Feedback On | Feedback Off
Serious Adverse Events (participants affected / at risk) | 0/815 | 0/771
Other Adverse Events (participants affected / at risk) | 0/815 | 0/771

LIMITATIONS AND CAVEATS:
Open label study - providers not blinded to intervention. High rates of missing CPR process measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No